CLINICAL TRIAL: NCT00180089
Title: Efficacy and Safety of Orale Budesonide in the Prevention of Acute Gastrointestinal Graft-versus-host Disease Following Allogenic Stem Cell Transplantation
Brief Title: Budesonide for Prevention of Acute Gastrointestinal GVHD Following Allogenic Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Dr. Falk Pharma GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PROGAST
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia; Graft-Versus-Host Disease
Keywords: graft-versus-host disease; budesonide; stem cell transplantation
MeSH Terms: conditions — Leukemia; Graft vs Host Disease | interventions — Budesonide

INTERVENTIONS:
Drug: Budesonide

SUMMARY:
The purpose of this study is to determine whether orale budesonide is effective in the prevention of acute gastrointestinal graft-versus-host disease (GVHD) following allogenic stem cell transplantation.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether orale budesonide is effective in the prevention of acute gastrointestinal graft-versus-host disease (GVHD) following allogenic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* planned allogenic stem cell or bone marrow transplantation
* HLA identity (max. 1 mismatch)
* standard GVHD prophylaxis with cyclosporin A or tacrolimus combined with MTX, +/- ATG or Campath1H
* written informed consent

Exclusion Criteria:

* history of allogenic transplantation
* in vitro T-cell depleted transplant
* pretreatment with budesonide within the previous 4 weeks
* known intolerance to budesonide
* gastrointestinal infections
* portal hypertension
* concomitant infectious diseases
* liver cirrhosis, impaired liver function
* severe mental disorder
* lack of compliance
* drug or alcohol abuse
* pregnancy, lactation
* childbearing potential without effective contraception

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2004-01; Primary Completion 2009-03 (Actual); Study Completion 2010-01

PRIMARY OUTCOMES:
incidence of acute gastrointestinal (GI) GVHD in the active group versus placebo group

SECONDARY OUTCOMES:
safety
grade of acute GI GVHD
incidence of chronic GI GVHD
incidence of infectious complications
overall and disease-free survival 1 yr after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Miehlke, Prof., Principal Investigator — Medical Department I, Technical University Hospital, Dresden, Germany
Locations (1):
- Medical Department I, Technical University Hospital, Dresden, Germany

REFERENCES:
- [Derived] Schmelz R, Bornhauser M, Schetelig J, Kiani A, Platzbecker U, Schwanebeck U, Grahlert X, Uharek L, Aust D, Baretton G, Schwerdtfeger R, Hampe J, Greinwald R, Mueller R, Ehninger G, Miehlke S. Randomised, double-blind, placebo-controlled trial of oral budesonide for prophylaxis of acute intestinal graft-versus-host disease after allogeneic stem cell transplantation (PROGAST). BMC Gastroenterol. 2014 Nov 26;14:197. doi: 10.1186/s12876-014-0197-7. PMID 25425214